CLINICAL TRIAL: NCT07031778
Title: Efficacy of Topical Application of Simvastatin in Bone Regeneration
Brief Title: Topic Simvastatin for Bone Regeneration
Acronym: SM
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Francisco Javier Manzano-Moreno, PhD, DDS, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3904/CEIH/2023; 3904/CEIH/2023 (Other: Ethics Committee University of Granada)
Record Dates: First submitted 2025-05-23; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Dimensional Changes; Bone Density
Keywords: simvastatin; bone density; dimensional changes; cbct scan
MeSH Terms: interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- drug intervention: Gel SM (Experimental): 30 lower third molars in whose alveolus post-extraction we will place simvastatin gel at 1.2%.
  Interventions: Drug: Simvastatin
- Drug intervention: Sm + collagen sponge (Active Comparator): 30 lower third molars in whose alveolus post-extraction we will place a collagen sponge impregnated with saline solution containing 10 mg of simvastatin.
  Interventions: Drug: Simvastatin 10 mg
- Control (Placebo Comparator): 30 lower third molars in whose alveolus post-extraction we will place a collagen sponge impregnated with gel without simvastatin
  Interventions: Drug: Simvastatin Placebo

INTERVENTIONS:
Drug: Simvastatin — Simvastatin gel with 1.2% simvastatin
  Arms: drug intervention: Gel SM
Drug: Simvastatin 10 mg — sponge of collagen impregned in saline solution with 10 mg of simvastatin
  Arms: Drug intervention: Sm + collagen sponge
Drug: Simvastatin Placebo — Collagen sponge impregned in simvastatin placebo gel without simvastatin
  Arms: Control

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of topical application of simvastatin in bone regeneration in the maxillae, in the reduction of dimensional bone changes, using mandibular third molar surgery as a model and assessing bone healing at 12 weeks. We will also compare the two forms of intralveolar topical administration currently used to assess which is the best form of administration. The main questions it aims to answer are:

* Can the topical application of simvastatin, used as a preservation material, improve the variations with respect to bone dimensions and density that occur after tooth extraction.
* Can topical application of SM improve soft tissue healing.
* Does the topical application of SM produce changes with respect to postoperative variables of pain, inflammation or trismus.
* What is the best vehicle for topical SM administration?

For this purpose, the investigators will randomly place 4 topical treatment options in the postextraction alveoli:

* SM in gel form
* collagen sponge impregnated with saline solution containing 10 mg of SM
* collagen sponge with placebo gel. All patients will undergo postoperative CBCT, which will be repeated at 12 weeks.

In addition, inflammation, trismus and pain variables will be measured preoperatively, at 24 hours, 3 and 7 days.

DETAILED DESCRIPTION:
The study design is a double-blind randomized clinical trial (RCT). The study population consisted of patients referred to the Master's Degree in Oral Surgery and Implantology of the Faculty of Dentistry of the UGR (Granada) with an indication for surgical extraction of mandibular third molars.

A sample of 90 third molars will be used to establish a confidence level of 95% and a power of 90%. The sample will be divided into 3 groups of 30 each. Group I: 30 mandibular third molars in which gel with 1.2% simvastatin is used for healing. Group II: 30 mandibular third molars in which a collagen sponge impregnated with saline solution containing 10 mg of the active ingredient simvastatin is used for healing. Group III: 30 mandibular third molars in which a collagen sponge impregnated in gel without SM is used for healing.

SURGICAL PROCEDURE:

Extraction will be performed only of included mandibular third molars. For this purpose we will anesthetize the lower dental nerve, lingual nerve and buccal nerve using 4% articaine with epinephrine by means of the truncular technique.

The intervention will be performed by flap lifting, ostectomy with handpiece and round bur, or odontosection with turbine whenever the case requires it. The socket will be curetted and washed with physiological saline solution to ensure that no surgical debris remains. After this, we will proceed to place in the socket the combination of material chosen by randomization (simvastatin gel, gel without simvastatin, collagen sponge with simvastatin or only collagen sponge). Once the filling material has been placed, we will proceed to the primary closure of the wound with 3.0 silk. We will place a gauze with 0.20% chlorhexidine gel at the end of the extraction, for the patient to keep it for 30 minutes. We will indicate to the patient the appropriate postoperative care and we will prescribe 0.12% chlorhexidine mouthwash for rinsing after brushing. One week later, the patient will be seen to remove the suture.

Postoperative medication:

* Antibiotic treatment: amoxicillin 750 mg 1 every 8 hours, for 7 days. In case of allergy to penicillin, the drug of choice will be clindamycin 300 mg 1 every 8 hours.
* Analgesic and anti-inflammatory treatment: ibuprofen 400 mg 1 every 8 hours for two days, from the third day on demand. Rescue paracetamol 1 g.

VARIABLES TO BE STUDIED

Primary Variables:

The primary variable to be studied will be the dimensional changes

Secondary variables:

The secondary variables to be studied will be bone density measured in Hounsfield units , soft tissue healing, pain and analgesia, inflammation and trismus.

ELIGIBILITY:
Inclusion Criteria:

* Anesthetic risk ASA I-II.
* Patients with the adjacent tooth in the mouth (37 or 47).
* Third molars with fully developed roots.
* Mandibular third molars included or semi-included.
* With indication for extraction.
* Signed informed consent.

Exclusion Criteria:

* Pregnant or lactating women.
* Chronic smokers.
* Patients with decompensated metabolic disease.
* Patients with motor difficulties that prevent or hinder hygiene.
* Patients who are using statins to treat hypercholesterolemia.
* Patients under treatment with drugs that could affect the osseointegration process such as chemotherapy drugs, bisphosphonates, corticosteroids or immunosuppressants.
* Patients with metabolic bone diseases or who have undergone radiotherapy in the last five years.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dimensional changes | From the time of extraction to when bone regeneration is supposed to be completed 12 weeks later.
  The primary variable to be studied will be the bone dimensional changes that occur after tooth extraction, both horizontally and vertically. These will be assessed by means of CBCT scans carried out immediately postoperatively (T0) and 12 weeks later (T1).

SECONDARY OUTCOMES:
Bone density | Postextraction to the end of bone regeneration at 12 week latter
  Bone density measured in Hounsfield units on CBCT post-extraction and at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- UGranada, Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Degala S, Bathija NA. Evaluation of the Efficacy of Simvastatin in Bone Regeneration after Surgical Removal of Bilaterally Impacted Third Molars-A Split-Mouth Randomized Clinical Trial. J Oral Maxillofac Surg. 2018 Sep;76(9):1847-1858. doi: 10.1016/j.joms.2018.04.035. Epub 2018 May 31. PMID 29859160
- [Background] Cruz R, Moraschini V, Calasans-Maia MD, de Almeida DCF, Sartoretto SC, Granjeiro JM. Clinical efficacy of simvastatin gel combined with polypropylene membrane on the healing of extraction sockets: A triple-blind, randomized clinical trial. Clin Oral Implants Res. 2021 Jun;32(6):711-720. doi: 10.1111/clr.13740. Epub 2021 Mar 27. PMID 33715258
- [Background] Deepanjali M, Prasad TS, Manodh P. Efficacy of simvastatin in bone regeneration after surgical removal of mandibular third molars. Oral Maxillofac Surg. 2023 Sep;27(3):427-432. doi: 10.1007/s10006-022-01081-y. Epub 2022 Jun 1. PMID 35648294
- [Background] Diniz JA, Barbirato DDS, do Nascimento EHL, Pontual ADA, Dourado ACAG, Laureano Filho JR. Tomographic evaluation of the effect of simvastatin topical use on alveolar bone microarchitecture, pain and swelling after mandibular third molar extraction: a randomized controlled trial. Clin Oral Investig. 2022 Apr;26(4):3533-3545. doi: 10.1007/s00784-021-04322-8. Epub 2022 Jan 22. PMID 35064813